CLINICAL TRIAL: NCT03328936
Title: Randomized Study of Personalized Melphalan Dosing in the Setting of Autologous Transplant
Brief Title: Study of Personalized Melphalan Dosing in the Setting of Autologous Transplant
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ashley Rosko, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU-17082; NCI-2017-01702 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA016058 (NIH)
Record Dates: First submitted 2017-10-03; First posted 2017-11-01 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Hematopoietic Cell Transplantation Recipient; Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (melphalan hydrochloride for 3-day severe neutropenia) (Experimental): Patients receive personalized dose of melphalan hydrochloride IV on day -2 for for predicted 3-day duration of severe neutropenia and undergo standard of care autologous stem cell transplant on day 0.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Melphalan Hydrochloride; Other: Pharmacological Study
- Arm II (melphalan hydrochloride or 5-day severe neutropenia)) (Experimental): Patients receive personalized dose of melphalan hydrochloride IV on day -2 for predicted 5-day duration of severe neutropenia and undergo standard of care autologous stem cell transplant on day 0.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Melphalan Hydrochloride; Other: Pharmacological Study

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Melphalan Hydrochloride — Given personalized dose IV for predicted 3-day duration of severe neutropenia
  Other Names: Alkeran; Alkerana; Evomela
  Arms: Arm I (melphalan hydrochloride for 3-day severe neutropenia)
Drug: Melphalan Hydrochloride — Given personalized dose IV for predicted 5-day duration of severe neutropenia
  Other Names: Alkeran; Alkerana; Evomela
  Arms: Arm II (melphalan hydrochloride or 5-day severe neutropenia))
Other: Pharmacological Study — Correlative studies

SUMMARY:
This randomized phase II trial studies the side effects and how well melphalan hydrochloride works in treating patients with multiple myeloma that has come back or does not respond to treatment. Drugs used in chemotherapy, such as melphalan hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Identify whether targeting approximate (approx.) 3- or 5-days of severe neutropenia after exposure to a personalized melphalan hydrochloride (melphalan) dose results in best clinical outcome.

II. Measure melphalan-related toxicities in both 3-day and 5-day arms. III. Measure response per International Myeloma Working Group (IMWG). IV. Record overall survival (OS) and progression free survival (PFS).

SECONDARY OBJECTIVES:

I. To administer a test dose of melphalan and obtain test dose melphalan pharmacokinetics (PK) data from the first 33 patients.

II. Measure drug-induced deoxyribonucleic acid (DNA) damage in peripheral blood mononuclear cells (PBMCs) treated with melphalan ex vivo post exposure.

III. Measure drug-induced DNA damage in patient myeloma cells treated with melphalan ex vivo.

IV. Assess melphalan-induced DNA damage in treated patients. V. Measure allele and genotype frequencies of variants, as well as gene expression of XRCC1 rs25487 and XRCC3 rs861529.

VI. Additional genetic variants relevant to DNA repair, melphalan transport, and clinical toxicities may be tested as well.

VII. Test cytotoxicity (half maximal inhibitory concentration [IC50]) of patient PBMCs prior to autologous transplant after exposure to melphalan ex vivo.

VIII. Measure p53 and phospho(TP53) in patient PBMCs prior to autologous transplant at baseline and after exposure to melphalan ex vivo.

IX. Incorporate both disease progression and drug-related toxicities into separate models linked to our calculated melphalan area under the curve (AUC) model.

OUTLINE: Patients are randomized into 1 of 2 arms.

ARM I: Patients receive personalized dose of melphalan hydrochloride intravenously (IV) on day -2 for predicted 3-day duration of severe neutropenia and undergo standard of care autologous stem cell transplant on day 0.

ARM II: Patients receive personalized dose of melphalan hydrochloride IV on day -2 for predicted 5-day duration of severe neutropenia and undergo standard of care autologous stem cell transplant on day 0.

After completion of study treatment, patients are followed up for 30 days, at 3 months after transplant, and then every 6-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have relapsed or refractory myeloma that fits or did fit IMWG diagnostic criteria for multiple myeloma; patients with AL amyloidosis and polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes (POEMS) are excluded; measurable disease is not required
* Patient undergoing autologous transplant as part of first line therapy
* All races and ethnic groups are eligible for this study
* Patients must also have an adequate autologous graft as defined as a cryopreserved peripheral blood stem cell (PBSC) graft containing > 2 x 10^6 CD34+ cells/kg patient weight
* Eastern Cooperative Oncology Group (ECOG) performance status < 2 (Karnofsky > 60%) is required for eligibility; those patients with lower performance status based solely on bone pain secondary to multiple myeloma are eligible
* Absolute neutrophil count (ANC) > 1000/uL
* Platelet count > 50,000
* Transfusion independent
* Total bilirubin < 1.5 mg/dL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 x the institutional upper limit of normal
* Left ventricular ejection fraction >= 40%
* Carbon monoxide diffusing capability (DLCO) > 50% predicted
* Forced expiratory volume in 1 second (FEV1) > 50% predicted
* Forced vital capacity (FVC) > 50% predicted
* Ability to understand and willingness to sign a written informed consent document
* Females of childbearing potential (FCBP) must not be pregnant as per institutional standard; if no institutional standard exists, then patients must have a negative serum or urine pregnancy test prior to transplant; a female of childbearing potential (FCBP) is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)

Exclusion Criteria:

* Patients who are receiving any other anti-myeloma investigational agents
* Uncontrolled illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, myocardial infarction in the preceding 6 months, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued
* Patients with a "currently active" second malignancy that, in the opinion of the principal investigator, will interfere with patient participation, increase patient risk, shorten survival to < 1 year, or confound data interpretation
* Concurrent use of complementary or alternative medicines that in the opinion of the principal investigator would confound the interpretation of toxicities and/or antitumor activity of the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Complete response proportion | At 90 days
  Complete response will be defined as complete response + stringent complete response according to the International Myeloma Working Group Uniform response criterion. Will be calculated with an exact 95% confidence interval, both within arms and across arms.

SECONDARY OUTCOMES:
Incidence of melphalan hydrochloride-related toxicities | Up to 3.5 years
  Will assess melphalan-related toxicities (possibly, probably, or definitely related to high dose melphalan) including the incidence of grade 3/4 mucositis, grade 3/4 bacteremia, length of inpatient stay, duration of severe neutropenia (absolute neutrophil count < 500), duration of severe thrombocytopenia (Platelet < 20K), and proportion with tachyarrhythmias (e.g. atrial fibrillation with rapid ventricular rate).
Minimal residual disease negative proportions | Pre-transplant
  Will be assessed by standard next generation sequencing.
Minimal residual disease negative proportions | up to 1 year
  Will be assessed by standard next generation sequencing.
Overall survival | time from randomization to death, assessed up to 3.5 years
  Will be assessed.
Progression free survival | Time from transplant to death, clinical relapse, progressive disease, and death in all treated patients, assessed up to 3.5 years
  Will be assessed.
Time to biochemical relapse | Time from start of melphalan hydrochloride until the earliest of the following time points: progressive disease, clinical relapse, or relapse from complete response, assessed up to 3.5 years
  Will be assessed.
Time to progression | Time from start of melphalan hydrochloride until the criteria for disease progression are met, assessed up to 3.5 years
  Will be assessed.

OTHER OUTCOMES:
Deoxyribonucleic acid (DNA) damage repair | Up to 3.5 years
  Will compare DNA damage repair efficiency in patients that have minimal response to induction and high dose melphalan hydrochloride (partial response or less) compared to those that are sequencing minimal residual disease negative.
Half maximal inhibitory concentration (IC50) | Up to 3.5 years
  Will create a multivariate linear regression model that includes each patient?s IC50, DNA repair gene single nucleotide polymorphism (SNP) presence or absence, and revised Multiple Myeloma International Staging System with progression free survival as the outcome.
Melphalan hydrochloride pharmacokinetics (PK) parameters | Within 2 hours prior to start of melphalan hydrochloride infusion and at 5, 30, 45, and 60 minutes, and 3 and 6 hours
  Will compare the prediction accuracy of melphalan hydrochloride pharmacokinetics using the test dose versus the current PK model. Test the use of aspects of test dose PK as a covariate in the current high dose melphalan hydrochloride prediction model.
p53 messenger ribonucleic acid | Up to 3.5 years
  Will correlate with progression free survival.
Phosphorylated TP53 | Up to 3.5 years
  Will correlate with progression free survival.
PK/pharmacodynamics (PD) model | Up to 3.5 years
  Will determine the parameter accuracy and precision of the newly integrated PK/PD model for absolute neutrophil count, mucositis, tachyarrhythmias, and disease progression.
XRCC1 rs25487 and XRCC3 rs861529 variant alleles | Up to 3.5 years
  Will use Cox survival analysis, measure progression free survival of patients with XRCC1 rs25487 and XRCC3 rs861529 variant alleles compared to wild type.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Rosko, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu